CLINICAL TRIAL: NCT02381197
Title: Diagnosis and Prediction of Preeclampsia: A Longitudinal Study of the Clinical Utility of Congo Red Dot Test in Bangladesh and Mexico
Brief Title: Longitudinal Study: Diagnosis and Prediction of Pre-Eclampsia by Using Congo Red Dot Test in Bangladesh and Mexico
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gynuity Health Projects (Other)
Collaborators: Nationwide Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 4004-B
Record Dates: First submitted 2015-02-25; First posted 2015-03-06 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Preeclampsia
Keywords: Congo Red Dot Test
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urine samples collected
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- pregnant women: Women presenting for prenatal care will provide urine samples at each antenatal care visit. The sample will be used to perform a Congo Red Dot test.
  Interventions: Device: Congo Red Dot test

INTERVENTIONS:
Device: Congo Red Dot test — The Congo Red Dot test is a simple dye test that detects unfolded or misfolded proteins

SUMMARY:
A population-based prospective cohort design will evaluate the progression of urine congophilia in pregnancy using the Congo Red Dot test by following patients longitudinally across gestation in Bangladesh and Mexico City.

DETAILED DESCRIPTION:
A population-based prospective cohort design will evaluate the progression of urine congophilia in pregnancy using the Congo Red Dot test by following patients longitudinally across gestation in Bangladesh and Mexico City. A total of 2000 women presenting for prenatal care will be enrolled (1000 at each site). In Bangladesh, pregnant women will be identified during monthly home visits of Community Health Workers (CHW) affiliated with Matlab in Chandpur and asked to participate. In Mexico, women will be identified at routine antenatal appointments. If the woman agrees to participate, investigators will ask her to consent to donation of urine for testing (Congo Red Dot test and Proteinuria dipstick test) at the time of enrollment, four times during her pregnancy (first trimester 6-12 weeks; second trimester 13-28 weeks; third trimester 29-36 weeks; term 37-41 weeks) and possibly three times postpartum (24 hours after delivery and daily until discharge). As a result, the enrolled patients will be followed longitudinally throughout pregnancy until delivery of the baby either at term for an uncomplicated gestation or preterm/term for preeclampsia. The group of women who develop preeclampsia will represent the study group. At the end of the study, the results will be analyzed to identify how many weeks in advance the women who developed preeclampsia displayed congophilia.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* Willing to give urine samples at prenatal visits
* Eligible to consent to research

Exclusion Criteria:

- None

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: In Bangladesh, pregnant women will be identified during monthly home visits of Community Health Workers (CHW) affiliated with Matlab in Chandpur and asked to participate. In Mexico, women will be identified at routine antenatal appointments at Hospital Materno-Infantil Inguarán.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Prevalence of urine congophilia | within 15 days of urine sample collection
  Use the Congo Red Dot test to identify urine congophilia among participants and evaluate progression of urine congophilia in pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Irina Buhimschi, Dr, Principal Investigator — Nationwide Children's Hospital; Beverly Winikoff, Dr, Principal Investigator — Gynuity Health Projects
Locations (2):
- Matlab, Chāndpur, Bangladesh
- Hospital Materno-Infantil Inguarán, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available to the public.